CLINICAL TRIAL: NCT00748878
Title: Platelet Function During ECMO
Brief Title: Platelet Function During ECMO (Extra Corporeal Membrane Oxygenation)
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Donald Null M.D., University of Utah / Primary Childrens Medical Center
Other Study IDs: 28645
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Platelet Function; Thrombocytopenia
Keywords: To better understand platelet function during ECMO
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Platelet transfusions are routinely administered during neonatal ECMO, with an average of 1.3 platelet transfusions per day being administered while a patient is undergoing ECMO treatment. The cause of thrombocytopenia during ECMO largely involves platelet adherence to the oxygenator membrane. Platelet transfusions carry risks such as infections with bacteria or yeast, and development or worsening of pulmonary hypertension. It is likely that if fewer platelet transfusions can be administered during the ECMO run, the cumulative adverse effects of platelet transfusions would diminish and patient outcomes improve. In order to better understand platelet function during ECMO, the investigators plan to serially determine the circulating platelet mass, plasma platelet factor 4 concentration, megakaryocyte mass (estimated by plasma thrombopoietin concentration), and platelet function as quantified by PFA100. Any patient on ECMO will be eligible for this pilot study of 5 patients. By understanding changes in platelet function, we hope to design a future study that may modify the frequency or need for platelet transfusions during ECMO.

DETAILED DESCRIPTION:
Platelet transfusions are routinely administered during neonatal ECMO, with an average of 1.3 platelet transfusions per day being administered while a patient is undergoing ECMO treatment.1 In general, a platelet transfusion is ordered for a patient on ECMO if the platelet count falls below 100,000/uL in order to prevent generalized hemorrhaging.1,2 The cause of thrombocytopenia during ECMO largely involves platelet adherence to the oxygenator membrane,3 but other mechanisms are also likely to be involved.4 Platelet transfusions carry risks as well as benefits.5 Infections with bacteria or yeast are the most commonly reported complications of platelet transfusions,6,7 but with multiple platelet transfusions the development or worsening of pulmonary hypertension may be another common adverse effect.8,9 Pulmonary hypertension can be the result of administering biologically active pro-inflammatory proteins (known to be present in platelet transfusions) into the venous circulation. Of note, the first capillary bed encountered will be within the pulmonary circulation.

It is likely that if fewer platelet transfusions could safely be administered during the ECMO run, the cumulative adverse effects of platelet transfusions would diminish and thereby patient outcomes might improve.

ELIGIBILITY:
Inclusion Criteria:

* Any patient on ECMO will be eligible for study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient on ECMO will be eligible for study.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2008-06; Primary Completion 2012-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald .Null, M.D., Principal Investigator — University of Utah
Locations (1):
- Primary Children's Medical Center, Salt Lake City, Utah, United States